CLINICAL TRIAL: NCT02425124
Title: Strengthening Mental Health Care in Chronic Care Patients With Hypertension. A Cluster Randomised Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of KwaZulu (Other)
Collaborators: Department for International Development, United Kingdom (Other Government); University of Cape Town (Other); King's College London (Other)
Responsible Party: Principal Investigator, Inge Petersen, Professor, University of KwaZulu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HRPC10
Record Dates: First submitted 2015-04-10; First posted 2015-04-23 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Depression; Hypertension
MeSH Terms: conditions — Depression; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): PC101 Enhanced usual primary health care where non-physician clinicians have been equipped with the basic skills to identify stress and depression/anxiety but with limited access to doctors authorized to prescribe antidepressant medication, and with no specific psychosocial interventions.
  Interventions: Behavioral: PC101+Mental Health
- Intervention (Experimental): PC101 + Mental Health Facility-based stepped care intervention combining stress and depression case detection and management by non-physician clinicians and referral pathways for anti-depressant medication and/or group/individual counselling delivered by lay-health workers for patients with depression.
  Interventions: Behavioral: PC101+Mental Health

INTERVENTIONS:
Behavioral: PC101+Mental Health — Facility-based stepped care intervention combining stress and depression case detection and management by non-physician clinicians and referral pathways for anti-depressant medication and/or group/individual counselling delivered by lay-health workers for patients with depression.

SUMMARY:
A pragmatic cluster randomized controlled trial (RCT) in 20 public sector primary care clinics in the Dr Kenneth Kaunda district of the North West Province of South Africa to assess mental health and health outcomes for depressed adults receiving hypertensive treatment by measuring the real-world effectiveness of a facility-based stepped care intervention combining stress and depression case detection and management by non-physician clinicians and referral pathways for anti-depressant medication and/or group/individual counselling delivered by lay-health workers for patients with depression. The control condition is enhanced usual primary health care where non-physician clinicians have been equipped with the basic skills to identify stress and depression/anxiety but with limited access to doctors authorized to prescribe antidepressant medication, and with no specific psychosocial interventions.

DETAILED DESCRIPTION:
Cardiovascular disease (hypertension and stroke) is the leading cause of mortality in the world and the second leading cause of death in Africa. Estimates by the WHO using disability adjusted life years (DALYs) suggest that NCDs were responsible for 28% of the total burden of disease in South Africa in 2004, with heart disease, diabetes and stroke together being responsible for the second most important cause of death in adult South Africans. In the investigators 2014 survey of 3 primary health care facilities in the North West Province where the Department of Health is piloting Integrated Chronic Disease Management the investigators found that of the 1 250 chronic care patients surveyed, 51% reported having hypertension. Spurring the rising burden of NCDs are mental disorders. One in 6 adults experience a common mental disorder (depression, anxiety disorders and substance use disorders) within a 12 month period (Herman et al., 2009), one in four receive treatment of any kind (Seedat et al., 2009). Depression co-exists with NCDs having a mutually reinforcing relationship compromising both prevention and treatment through exacerbating modifiable risk factors and compromising adherence and self-care respectively. Objectives: The investigators propose to strengthen the Primary Care 101 guidelines. This is a set of clinical guidelines and decision support for nurses developed for the identification and management of multiple chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

Clinics

* Twenty (20) largest clinics providing chronic care Patients
* Receiving hypertensive treatment at time of enrolment
* Depressive symptoms as indicated by total score of 9 or more on PHQ-9
* Planning to reside in area for the next year
* Capable of actively engaging in interviewer-administered questionnaire at time of recruitment, 6 months and 12 months later
* Written consent to participate in the study

Exclusion Criteria:

Clinics

* Clinics that do not provide Integrated Chronic Disease Management
* Small (<10 000 attendances/ year)
* Mobile or satellite
* Participated in piloting of intervention & data collection. Patients
* Inability to meet the above inclusion criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1052 (Actual)
Dates: Start 2015-04-22 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Depression | 6 Months
  50 % reduction in PHQ-9 score

SECONDARY OUTCOMES:
Depression | 12 months
  50 % reduction in the PHQ-9 score
Depression | 12 months
  Remission defined as score of <5 on PHQ9
Depression | 6 months; 12 months
  Mean PHQ9 scores
Blood pressure | 6 months and 12 months
  Difference in means
Disability | 12 Months
  Mean score using the Manual for WHO Disability Schedule WHODAS 2.0 schedule
Stress | 12 Months
  Mean score using Perceived Stress Scale
Antidepressant treatment | 12 months
  Proportion with antidepressant treatment initiated or intensified
Counselling | 12 months
  Proportion receiving counselling by clinic-based counsellor
Referral to specialist mental health worker/service | 12 months
  Proportion referred
Retention in care | 12 months
  Proportion in care
Cardiovascular risk factors | 12 months
  Difference in means
Diagnosis of other comorbid illnesses | 12 months
  Proportion diagnosed
Quality of chronic illness care received | 12 months
  Mean Patient Assessment of Care for Chronic Conditions (PACIC) score
Healthcare utilization | 12 months
  Incidence rate ratio using linkage with hospitalisation databases
Productivity and economic outcomes | 12 months
  Productivity and economic outcomes
All cause mortality | 12 months
  Proportion died

CONTACTS AND LOCATIONS:
Overall Officials: Inge Petersen, PhD, Principal Investigator — University of KwaZulu; Lara R Fairall, PhD, Principal Investigator — University of Cape Town; Graham Thornicroft, PhD, Principal Investigator — King's College London
Locations (1):
- Primary Health Care Facilities, Dr Kenneth Kaunda District, North West, South Africa

REFERENCES:
- [Derived] Petersen I, Fairall L, Zani B, Bhana A, Lombard C, Folb N, Selohilwe O, Georgeu-Pepper D, Petrus R, Mntambo N, Kathree T, Bachmann M, Levitt N, Thornicroft G, Lund C. Effectiveness of a task-sharing collaborative care model for identification and management of depressive symptoms in patients with hypertension attending public sector primary care clinics in South Africa: pragmatic parallel cluster randomised controlled trial. J Affect Disord. 2021 Mar 1;282:112-121. doi: 10.1016/j.jad.2020.12.123. Epub 2020 Dec 28. PMID 33412490
- [Derived] Petersen I, Bhana A, Folb N, Thornicroft G, Zani B, Selohilwe O, Petrus R, Mntambo N, Georgeu-Pepper D, Kathree T, Lund C, Lombard C, Bachmann M, Gaziano T, Levitt N, Fairall L; PRIME-SA research team. Collaborative care for the detection and management of depression among adults with hypertension in South Africa: study protocol for the PRIME-SA randomised controlled trial. Trials. 2018 Mar 22;19(1):192. doi: 10.1186/s13063-018-2518-6. PMID 29566730